CLINICAL TRIAL: NCT01611922
Title: Optimization of Assessment and Grading for Lid Wiper Epitheliopathy
Acronym: BURNABY
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: P/365/11/L
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Dry Eye
Keywords: eye; eyelid; contact lenses; dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Fluorescein; Contact Lenses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Symptomatic Lens Wearers: Contact lens wearers reporting a habitual wear time of less than eight hours and a noticeable reduction in comfort over a wearing day
  Interventions: Other: Ophthalmic dye; Device: Contact lenses
- Non-Symptomatic Contact Lens Wearers: Contact lens wearers reporting a comfortable wear time of more than 10 hours and minimal reduction in comfort over a wearing day
  Interventions: Other: Ophthalmic dye; Device: Contact lenses
- Asymptomatic Non-Contact Lens Wearers: Non-contact lens wearers reporting a minimal reduction in ocular comfort over the course of a day
  Interventions: Other: Ophthalmic dye

INTERVENTIONS:
Other: Ophthalmic dye — Topically instilled for the purpose of assessing lid margin staining
  Other Names: Lissamine Green; Sodium Fluorescein
Device: Contact lenses — Silicone hydrogel contact lenses per subject's habitual brand and power, worn for a minimum of 8 hours on the day of assessment, after which lenses will be removed and dye will be instilled.
  Groups: Non-Symptomatic Contact Lens Wearers; Symptomatic Lens Wearers

SUMMARY:
The purpose of this study is to assess eyelid margin staining, termed "lid wiper epitheliopathy" (LWE), in three populations. The hypothesis is LWE will be more prevalent in symptomatic contact lens wearers than non-symptomatic contact lens wearers and least prevalent in asymptomatic non-contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Has had an ocular examination in the last two years;
* Has clear corneas and no active ocular disease;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Has any ocular disease;
* Has a systemic condition that may affect a study outcome variable;
* Is using any systemic or topical medications that may affect ocular health;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Has undergone corneal refractive surgery;
* Currently wears contact lenses on an extended wear basis (overnight);
* Has any clinically significant lid or conjunctival abnormalities, neovascularization, corneal scars or corneal opacities;
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified and screened by the University of Waterloo in Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
LWE-associated staining score | 3 minutes after dye instillation
  Lens wearers must wear lenses for a minimum of 8 hours on the day of assessment, after which lenses will be removed and dye will be instilled. LWE-associated staining will be assessed by the investigator and reported as a composite score based on Korb's method.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, FCOptom, PhD, Principal Investigator — Centre for Contact Lens Research, School of Optometry, University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Canada